CLINICAL TRIAL: NCT05981404
Title: Impact of ß-glucan Supplementation During Calorie and Carbohydrate Restriction on Subjective Appetite and Gastrointestinal Appetite Hormones in Overweight Adults.
Brief Title: Impact of ß-glucan Supplementation on Subjective Appetite and Gastrointestinal Appetite Hormones.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Dalia Malkova, Coordinator of L4 Nutrition Programmes, Senior Lecturer., University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 200210051
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Experimental trial beta-glucan or experimental trial control (placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low calorie and low carbohydrate meals with β-glucan. (Experimental): On day 1, a low-calorie breakfast will be consumed at the metabolic investigation laboratory at New Lister Building (NLB) of Glasgow Royal Infirmary but low carbohydrate lunch and low-calorie dinner at home. On day 2, breakfast and lunch will be consumed at the laboratory and, prior to the breakfast, 1000mg of paracetamol will be taken, blood samples, breath hydrogen tests, appetite questionnaires will be obtained for 7 hours after the completion of breakfast. 3g β-glucan will be consumed with each meal on both days.
  Interventions: Dietary Supplement: β-glucan
- Low calorie and low carbohydrate meals with placebo. (Experimental): On day 1, a low-calorie breakfast will be consumed at the metabolic investigation laboratory at New Lister Building (NLB) of Glasgow Royal Infirmary but low carbohydrate lunch and low-calorie dinner at home. On day 2, breakfast and lunch will be consumed at the laboratory and, prior to the breakfast, 1000mg of paracetamol will be taken, blood samples, breath hydrogen tests, appetite questionnaires will be obtained for 7 hours after the completion of breakfast. 3g cellulose will be consumed with each meal on both days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: β-glucan — Consuming 3g β-glucan with each meal.
  Arms: Low calorie and low carbohydrate meals with β-glucan.
Dietary Supplement: Placebo — Consuming 3g Cellulose with each meal.
  Arms: Low calorie and low carbohydrate meals with placebo.

SUMMARY:
The goal of this clinical trial is to how supplementation with beta -glucan during two days of caloric and carbohydrate restriction impacts subjective appetite and gastrointestinal appetite hormones in healthy overweight adults. In addition, the study aims to investigate the impact on gastric emptying since appetite and energy intake following food or supplement consumption can also relate to their impact on gastric emptying and as reduced hunger and enhanced satiety have been reported to be linked with delayed gastric emptying. The study will also investigate how these interactions impact after meal responses of insulin and glucose and thus insulin sensitivity. The caloric restriction during breakfasts and dinners will be achieved by low-calorie ready meals in the format of the counterweight PRO800 diet and lunches will be low in carbohydrates. It aims to test whether the addition of β-glucan to calorie and carbohydrate-restricted meals amends postprandial responses of appetite hormones and subjective appetite.

participated will be assigned in double-blinded randomised crossover study, intervention group will be supplemented with 3g beta-glucan and the control group supplemented with 3g placebo.

DETAILED DESCRIPTION:
This will be a randomised crossover study which will be conducted on overweight and obese women with BMI of 27-35 kg/m2 and 18 -50 years old. Subjects will conduct two experimental trials, each lasting over 2 days and involving the consumption of two low-calorie meal replacements, one for breakfast and another one for dinner, and a low carbohydrate lunch meal for 2 consecutive days. In one trial, during each meal participants will take 3g of beta-glucan supplement and 3 g of cellulose as a placebo will be taken in another trial. On day 1 of each trial, a low-calorie breakfast will be consumed at the metabolic investigation laboratory at New Lister Building (NLB) of Glasgow Royal Infirmary and low carbohydrate lunch and low-calorie dinner at home. On day 2, breakfast and lunch will be consumed at the laboratory. On day 2, prior to the breakfast, 1000mg of paracetamol will be taken, and blood samples, breath hydrogen tests, appetite questionnaires and metabolic rate measurements will be obtained for 7 hours after the completion of breakfast. Trials will be separated by a 7-day washout period. All measurements will be collected at New Lister Building (NLB). Prior to the main experimental trials, participants will be asked to undergo a screening session which includes answering a health screening questionnaire and undergoing measurements of height, body weight, body composition and resting energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

Participants will be asked to confirm whether they had stable body weight for at least 3 months and are not following a diet to gain or lose weight. They will also be asked to confirm that they are non-smokers, not on long-term medication, not pregnant or lactating, and have no known food allergies to the ingredients in test meals and to Paracetamol.

Exclusion Criteria:

Participants will be excluded if they are smokers and have irregular menstruation cycles, use any type of medication, exercised more than 75min a week, were pregnant or lactating. Participants will be required to be free of any medical condition, including having food allergies and stable body weight for at least 3 months preceding the study. Participants will be excluded if they are allergic to paracetamol and any types of food and were following any weight loss diet for the last 3 months, are vegan or vegetarian or follow any diet other than the typical Western diet. Participants will be expected to be not on any kind of dietary supplement at the time of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in gastrointestinal appetite hormones and appetite scores between the two groups. | On day 2 of each experimental trial.
  Taking blood samples every 30 minutes to test the changes in appetite hormones. Asking participants to answer questionnaires which will be calculated by Validated Visual Analogue Scale (VAS). The scale is 100 mm in length with words anchored to a minimum and a maximum of the ''desire to eat'', ''fullness'', ''hunger'' and ''satiety'' the point corresponding to their sensations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fechner E, Smeets ETHC, Schrauwen P, Mensink RP. The Effects of Different Degrees of Carbohydrate Restriction and Carbohydrate Replacement on Cardiometabolic Risk Markers in Humans-A Systematic Review and Meta-Analysis. Nutrients. 2020 Apr 2;12(4):991. doi: 10.3390/nu12040991. PMID 32252374
- [Result] Wang GJ, Tomasi D, Backus W, Wang R, Telang F, Geliebter A, Korner J, Bauman A, Fowler JS, Thanos PK, Volkow ND. Gastric distention activates satiety circuitry in the human brain. Neuroimage. 2008 Feb 15;39(4):1824-31. doi: 10.1016/j.neuroimage.2007.11.008. Epub 2007 Nov 22. PMID 18155924
- [Result] Thom G, Dombrowski SU, Brosnahan N, Algindan YY, Rosario Lopez-Gonzalez M, Roditi G, Lean MEJ, Malkova D. The role of appetite-related hormones, adaptive thermogenesis, perceived hunger and stress in long-term weight-loss maintenance: a mixed-methods study. Eur J Clin Nutr. 2020 Apr;74(4):622-632. doi: 10.1038/s41430-020-0568-9. Epub 2020 Feb 4. PMID 32020057
- [Result] Miyamoto J, Watanabe K, Taira S, Kasubuchi M, Li X, Irie J, Itoh H, Kimura I. Barley beta-glucan improves metabolic condition via short-chain fatty acids produced by gut microbial fermentation in high fat diet fed mice. PLoS One. 2018 Apr 26;13(4):e0196579. doi: 10.1371/journal.pone.0196579. eCollection 2018. PMID 29698465
- [Result] Ebbeling CB, Feldman HA, Klein GL, Wong JMW, Bielak L, Steltz SK, Luoto PK, Wolfe RR, Wong WW, Ludwig DS. Effects of a low carbohydrate diet on energy expenditure during weight loss maintenance: randomized trial. BMJ. 2018 Nov 14;363:k4583. doi: 10.1136/bmj.k4583. PMID 30429127